CLINICAL TRIAL: NCT06406088
Title: EarGenie Minimum Viable Product (MVP) Performance Evaluation: Sensitivity and Specificity of a Test of Sound Detection and Discrimination Using Functional Near-infrared Spectroscopy (fNIRS) in a Single Group Trial of Normal Hearing Infants
Brief Title: EarGenie MVP Performance Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Bionics Institute of Australia (Other)
Responsible Party: Principal Investigator, Colette McKay, Leader, Translational Hearing Research and Principal Scientist, The Bionics Institute of Australia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 105500
Record Dates: First submitted 2024-05-01; First posted 2024-05-09 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Hearing Impaired Children
Keywords: fNIRS

STUDY DESIGN:
Intervention Model Description: A single group of infants without hearing impairment will be recruited so that the performance of the two EarGenie MVP tests of speech sound detection and discrimination can be estimated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EarGenie MVP (Experimental): Infants who have a test completed with EarGenie MVP in a single test session
  Interventions: Device: EarGenie MVP test

INTERVENTIONS:
Device: EarGenie MVP test — The EarGenie MVP test consists of placing the EarGenie headgear containing light emitting diodes (LEDs) and light detectors on the infant and running the fNIRS tests of sound detection or sound discrimination via the user interface. Blocks of speech sounds are presented to the infant via earphones or via speaker, and the EarGenie MVP measures changes in the blood oxygenation in temporal and prefrontal regions of the cortex. Automatic analyses are run to determine whether the infant heard the sounds (at levels 35, 50, and 65 dBSPL) or discriminated between two sounds (Ba/Tea, Ba/Bee, or Ba/Ga). The infant will be in a natural sleep or quiet awake state when the fNIRS test is run. Prior to the test, standard audiometric procedures (otoscopy and tympanometry) will confirm normal middle ear function.

SUMMARY:
This is a single-group clinical trial to evaluate the performance of the EarGenie minimum viable product (MVP) in normal hearing infants. The EarGenie MVP tests for detection and discrimination of sounds will be administered, and the sensitivity and specificity of the tests will be estimated for a range of sound levels (detection) and speech sound contrasts (discrimination).

DETAILED DESCRIPTION:
Procedures:

All procedures will be carried out in a single test session.

Determination of infant eligibility will be undertaken by confirming that the infant has passed hearing screening or diagnostic audiological assessment and is under the age of 2 years.

Before completing the fNIRS tests, the infant will undergo otoscopy and tympanometry to exclude possible temporary conductive hearing loss associated with abnormal tympanometric results. These are standard audiological procedures. If the infant has abnormal tympanometric results in both ears on the day, the test session will be rescheduled. The parent/guardian will be advised of the finding and its possible consequences (possible conductive hearing loss, possible progression to acute otitis media) and advised to seek medical advice should the infant show signs of illness or if hearing loss is suspected.

All assessments in the fNIRS test session will be undertaken by qualified paediatric audiologists who are trained in the fNIRS procedures.

For the fNIRS tests, the infant will be asleep or in a quietly entertained response state.

After the headgear is placed on the infant's head, an optode calibration procedure is undertaken to ensure the equipment is ready. During the actual test, blocks of speech sounds lasting 5.4 seconds will be played to the infant either via tubephone or via speakers. During and after the test session, the infant will be monitored for any signs of discomfort or distress. Testing will discontinue if the infant is not either asleep or in a quiet response state.

For the detection test, a single speech sound "BA" will be presented at several levels (35, 50, and 65 dBSPL), and the test blocks will include "no sound" blocks to allow estimates of false positive results.

For the discrimination test, three different speech contrasts will be presented ("BA/TEA", "BA/BEE", and "BA/GA") at 65 dB SPL. The test will also include blocks of "BA/BA" to allow estimates of false positive rates.

For each infant, the sound levels at which "BA" evoked a statistically significant response will be recorded, and/or the speech contrasts which evoked a significant discrimination response will be recorded. Each infant will either have a detection test or a discrimination test, or both if their response state allows. At least 50 full detection and 50 full discrimination test results for estimating sensitivity and specificity outcome measures will be obtained.

ELIGIBILITY:
Inclusion Criteria:

Each infant must meet all of the following criteria to be enrolled in this trial:

* Is between the ages of 1 and 24 months at the time of fNIRS testing.
* Has no known hearing loss, having either passed newborn hearing screening or diagnostic audiological assessment.
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Exclusion Criteria:

* Infants with skin conditions such as cradle cap, eczema, or other skin conditions on the head will be excluded.

There are no additional exclusion criteria other than not meeting the inclusion criteria.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Performance of the EarGenie test of sound detection for a range of sound levels in normal-hearing infants. | Up to 18 months
  The primary outcome 1 is a set of test results that allow the sensitivity and specificity of the test to be estimated within +/-5% accuracy. Outcome measures (sensitivity and specificity) will be calculated for the detection test for three audible sound levels (65, 50, 35 dBSPL) within the comfortable loudness range.
  Sensitivity for the detection test will be estimated as the proportion of infants for whom the test result showed a positive detection and specificity will be estimated as [1- the proportion of infants whose test result for a control condition (silence) showed a (false) detection].
Performance of the EarGenie test of speech discrimination for a range of speech sound contrasts in normal-hearing infants | Up to 18 months
  The primary outcome 2 is a set of test results that allow the sensitivity and specificity of the test to be estimated within +/-5% accuracy. Outcome measures (sensitivity and specificity) will be calculated for the discrimination test for three difference speech sound contrasts differing in difficulty (BA/TEA, BA/BEE, and BA/GA), all presented at 65 dB SPL.

CONTACTS AND LOCATIONS:
Overall Officials: Colette McKay, PhD, Principal Investigator — The Bionics Institute of Australia
Locations (1):
- Bionics Institute, Fitzroy, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No